CLINICAL TRIAL: NCT04854954
Title: Prediction of Secondary Neurological Deterioration in Patients With Moderate Traumatic Brain Injury : an Observational Study
Brief Title: Prediction of Secondary Neurological Deterioration in Patients With Moderate Traumatic Brain Injury
Acronym: PREDICT-TCM
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: PREDICT-TCM (29BRC20. 0136)
Record Dates: First submitted 2021-04-19; First posted 2021-04-22 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-01

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with moderate traumatic brain injury (mTBI) are 1,5 times more frequent than those with severe TBI and some of them will develop secondary neurologic deterioration (SND) within the first 7 days. However, identifying at risk patients of SND is still challenging. This study aimed to determine risk factors associated with SND after mTBI.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Admitted in Brest hospital between 2015 and 2018 for moderate TBI, defined by Glasgow coma scale (GCS) score 9-13

Exclusion Criteria:

* Non consenting patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults admitted in Brest hospital (ICU and wards) between 2015 and 2018 for moderate TB
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2021-03-22 (Actual)

PRIMARY OUTCOMES:
Secondary neurologic deterioration | Within 7 days after hospital admission
  SND was defined either by a decrease in GCS or by a deterioration in neurologic status sufficient to warrant intervention like mechanical ventilation, transfer to the ICU or neurosurgical intervention

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three months and ending five years following the publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement

REFERENCES:
- [Derived] Aries P, Ognard J, Cadieu A, Degos V, Huet O. Secondary Neurologic Deterioration After Moderate Traumatic Brain Injury: Development of a Multivariable Prediction Model and Proposition of a Simple Triage Score. Anesth Analg. 2024 Jan 1;138(1):171-179. doi: 10.1213/ANE.0000000000006460. Epub 2023 Apr 25. PMID 37097898